CLINICAL TRIAL: NCT07360197
Title: The Effect of Mindfulness-Based Stress Reduction Training on Fear of Childbirth and Psychological Well-being in Women Experiencing Premenstrual Syndrome
Brief Title: MBSR for Premenstrual Syndrome and Childbirth Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aysel AKBENIZ (Other)
Responsible Party: Sponsor-Investigator, Aysel AKBENIZ, Associate Professor of Psychiatric Nursing, Tarsus University
Organization: Tarsus University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INONU-CT-4615-MBSR
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Premenstrual Syndrome; Fear of Childbirth; Psychological Well-being
Keywords: Mindfulness-Based Stress Reduction; MBSR; Premenstrual Syndrome; Childbirth Fear; Psychological Well-being; Women's Mental Health; Behavioral Intervention; Randomized Controlled Trial
MeSH Terms: conditions — Premenstrual Syndrome; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR Intervention Group (Experimental): articipants in this arm received an 8-session Mindfulness-Based Stress Reduction (MBSR) program delivered online. Each session lasted 40 minutes and was conducted twice weekly. The program included mindfulness practices such as body scan, breath awareness, emotional awareness, and mindfulness-based coping strategies, along with home practice assignments.
  Interventions: Behavioral: MBSR Intervention Group
- Control Group (No Intervention): Participants in this arm did not receive any active intervention during the study period. They completed baseline and post-intervention assessments only and were provided with an information booklet after completion of the study.

INTERVENTIONS:
Behavioral: MBSR Intervention Group — A structured 8-session mindfulness-based stress reduction program designed to enhance awareness, emotion regulation, and stress coping. The intervention included guided mindfulness practices such as body scan, breathing exercises, emotional awareness, and cognitive mindfulness strategies delivered online by a certified instructor.
  Arms: MBSR Intervention Group

SUMMARY:
This randomized controlled trial evaluates the effectiveness of a Mindfulness-Based Stress Reduction (MBSR) program on premenstrual symptom severity, fear of childbirth, and psychological well-being in women experiencing Premenstrual Syndrome (PMS). PMS is a prevalent condition characterized by emotional, cognitive, and physical symptoms that significantly impair women's daily functioning, stress tolerance, and quality of life. In addition to its somatic and affective burden, PMS is associated with increased anxiety and emotional dysregulation, which may contribute to elevated fear related to pregnancy and childbirth during the preconception period.

A total of 126 women aged 18 years and older who met the diagnostic threshold for PMS (Premenstrual Syndrome Scale score ≥ 110) were enrolled between June 2023 and November 2025 and randomly assigned in a 1:1 ratio to either an MBSR intervention group or a control group. The intervention group received an eight-session online MBSR program delivered twice weekly, with each session lasting 40 minutes. The program included mindfulness-based practices such as body scan, breath awareness, emotion-focused mindfulness, and cognitive awareness exercises, supported by structured home practice assignments. The control group received no active intervention during the study period.

Primary and secondary outcomes were assessed using validated self-report instruments at baseline and after completion of the 8-week intervention period. Premenstrual symptom severity was measured using the Premenstrual Syndrome Scale (PMSS), fear of childbirth was evaluated with the Childbirth Fear-Prior to Pregnancy Scale (CF-PPS), and psychological well-being was assessed using the Psychological Well-Being Scale (PWBS).

The primary objective of the study is to determine whether participation in the MBSR program leads to a greater reduction in premenstrual symptom severity compared to a control condition. Secondary objectives include evaluating the effect of MBSR on reducing fear of childbirth and improving psychological well-being. This study aims to provide evidence for the effectiveness of a non-pharmacological, mindfulness-based intervention in supporting women's mental and reproductive health during the premenstrual period.

DETAILED DESCRIPTION:
Premenstrual Syndrome (PMS) is a common cyclical condition characterized by a wide range of physical, emotional, and behavioral symptoms that occur during the late luteal phase of the menstrual cycle. These symptoms, which include depressed mood, anxiety, irritability, fatigue, pain, and somatic discomfort, can significantly impair daily functioning, interpersonal relationships, academic and occupational performance, and overall quality of life. Beyond its somatic manifestations, PMS is increasingly recognized as a condition with substantial psychological and emotional consequences. Elevated stress reactivity, emotional dysregulation, and negative cognitive appraisals commonly observed in women with PMS may also contribute to heightened vulnerability to anxiety-related conditions, including fear of pregnancy and childbirth during the preconception period.

Fear of childbirth is a multidimensional construct encompassing cognitive, emotional, and physiological components, including catastrophic thinking, loss of control, bodily hypervigilance, and intolerance of uncertainty. Although most studies focus on fear of childbirth during pregnancy, emerging evidence suggests that such fear can develop long before conception, particularly among women experiencing high levels of anxiety, stress, and mood instability. Given the emotional and neuroendocrine fluctuations associated with PMS, women with severe premenstrual symptoms may be at increased risk for elevated fear related to pregnancy and childbirth. PMS has also been shown to negatively affect psychological well-being by reducing individuals' perceived sense of competence, life satisfaction, and capacity to cope with stress.

Mindfulness-Based Stress Reduction (MBSR) is a structured psychosocial intervention designed to enhance present-moment awareness, emotional regulation, and adaptive coping through mindfulness meditation, body awareness, and cognitive decentering. MBSR has demonstrated beneficial effects on stress, anxiety, depression, and psychological well-being in diverse clinical and non-clinical populations. By fostering nonjudgmental awareness of bodily sensations, emotions, and thoughts, MBSR may reduce the intensity of premenstrual symptoms, weaken maladaptive cognitive responses to discomfort, and improve overall psychological functioning. Furthermore, by promoting acceptance, self-regulation, and resilience, mindfulness-based approaches may reduce fear-related cognitive and emotional reactions associated with childbirth.

This study was designed as a randomized controlled trial to evaluate the effects of an MBSR program on premenstrual symptom severity, fear of childbirth, and psychological well-being in women experiencing PMS. The trial was conducted between June 2023 and November 2025. Eligible participants were women aged 18 years or older with regular menstrual cycles who met the diagnostic threshold for PMS based on a Premenstrual Syndrome Scale score of 110 or higher. Women with gynecological disorders or those using hormonal contraceptives were excluded.

After providing informed consent and completing baseline assessments, participants were randomly assigned in a 1:1 ratio to either the MBSR intervention group or a control group using computer-generated randomization. The intervention group received an eight-session MBSR program delivered online via Zoom. Sessions were conducted twice weekly, each lasting 40 minutes, and were facilitated by a certified mindfulness instructor. The program included structured mindfulness practices such as body scan, breath awareness, raisin exercise, attention to thoughts and emotions, and mindfulness-based coping strategies. Participants were encouraged to engage in regular home practice through assigned exercises. The control group did not receive any active intervention during the study period but completed the same assessment schedule.

Primary and secondary outcome measures were administered at baseline and immediately after completion of the 8-week intervention. Premenstrual symptom severity was assessed using the Premenstrual Syndrome Scale (PMSS), which evaluates emotional, cognitive, and somatic symptoms. Fear of childbirth was measured with the Childbirth Fear-Prior to Pregnancy Scale (CF-PPS), a validated instrument assessing fear related to pregnancy and birth before conception. Psychological well-being was evaluated using the Psychological Well-Being Scale (PWBS), which captures individuals' psychological resources, positive functioning, and overall mental well-being.

The primary objective of the study is to determine whether the MBSR intervention results in a greater reduction in PMS symptom severity compared with a control condition. Secondary objectives include assessing whether MBSR reduces fear of childbirth and enhances psychological well-being. Statistical analyses compare post-intervention outcomes between groups while controlling for baseline scores to estimate the effect of the intervention.

This trial aims to provide evidence for the role of mindfulness-based interventions as safe, feasible, and effective non-pharmacological strategies for improving women's mental health and reproductive well-being during the premenstrual period.

ELIGIBILITY:
Inclusion Criteria:

Female participants aged 18 years or older

Regular menstrual cycles (21-35 days)

Premenstrual Syndrome Scale (PMSS) total score ≥110

Willingness to participate and provide informed consent

Exclusion Criteria:

Presence of any gynecological disorder (e.g., abnormal uterine bleeding, fibroids, ovarian cysts)

Use of hormonal contraceptives or contraceptive pills

Failure to attend more than two MBSR sessions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Premenstrual Syndrome Severity | Baseline to 8 weeks
  Change in total score of the Premenstrual Syndrome Scale (PMSS) from baseline to post-intervention at 8 weeks.

SECONDARY OUTCOMES:
Fear of Childbirth | Baseline to 8 weeks
  Change in score on the Childbirth Fear - Prior to Pregnancy Scale (CF-PPS) from baseline to post-intervention at 8 weeks.
Psychological Well-being | Baseline to 8 weeks
  Change in total score on the Psychological Well-being Scale (PWBS) from baseline to post-intervention at 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No